CLINICAL TRIAL: NCT02942420
Title: Phase 2 Multi-Center, Dose Escalation Trial To Assess The Safety And Effectiveness Of Bucillamine On Urinary Cystine Excretion And Cystine Capacity In Patients With Cystinuria
Brief Title: Bucillamine Phase 2 Trial in Patients With Cystinuria
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Revive Therapeutics, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: REV401
Record Dates: First submitted 2016-10-19; First posted 2016-10-24 (Estimated); Last update posted 2017-05-18 (Actual); Status verified 2017-03

CONDITIONS: Cystinuria
MeSH Terms: conditions — Cystinuria | interventions — bucillamine

STUDY DESIGN:
Intervention Model Description: Dosing will occur sequentially from low to high dose: The 600 mg bucillamine dose group (Arm A) will enroll first, then after safety is assured, the 900 mg bucillamine dose group will enroll.
Masking Description: The study is unmasked, i.e., is open label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Group A (Experimental): Bucillamine 300 mg/day
  Interventions: Drug: Bucillamine
- Dose Group B (Experimental): Bucillamine 600 mg/day
  Interventions: Drug: Bucillamine

INTERVENTIONS:
Drug: Bucillamine — Thiol donor which results in a cysteine-bucillamine complex for removing excess cysteine from the urine

SUMMARY:
Subjects on a standard regimen of tiopronin (cystine binding thiol drug; CBTD) plus prescribed first-line therapy (i.e. on a hydration, alkali therapy and dietary restriction) who are failing therapy will be selected for this trial.

After completing informed consent, the subject will have Screening consisting of medication history and physical examination with vital signs. Samples of blood and urine will be taken for clinical laboratory and urinalysis. Patients will undergo a 12-lead ECG test. A history of side effects with current CBTD as well as laboratory recordings of abnormalities attributable to treatment will also be recorded.

Subjects will be dosed in a sequential manner, starting with the low dose group (300 mg/day), then proceeding to the 600 mg.day dose group.. Safety and tolerability will be monitored closely by an Independent Medical Monitor (IMM) and based on the IMM's assessment that it is safe to proceed to the higher dose (600 mg/day), subsequent subjects will be enrolled into that group. Up to 15 subjects each will be enrolled into either Group A or Group B.

After 7 days on the assigned bucillamine dose, a 24-hour urine sample will be taken and after completing the Day 8 safety visit, subjects will undergo a 7 day washout where no CBTDs will be taken. Thereafter, subjects will be allowed to resume their originally prescribed CBTDs under Investigator's supervision.

One week following study drug discontinuation, subjects will return to the clinic for follow-up safety assessments.

DETAILED DESCRIPTION:
Subjects on a standard regimen of tiopronin (cystine binding thiol drug; CBTD) plus prescribed first-line therapy (i.e. on a hydration, alkali therapy and dietary restriction) who are failing therapy will be selected for this trial.

Subjects will be encouraged to continue their usual self-selected ad-lib diets, fluid and alkali regimen and keep this regimen consistent throughout the duration of the study. Study diaries will be kept to assess consistency and drug compliance.

After completing informed consent, the enrolled subject will have an initial Screening interview. During the interview the patient will be assessed for symptoms of renal colic as well as asked about any scheduled urological procedures (a positive indication is an exclusionary criteria). At the Screening visit, a medication history will be taken and a complete physical examination, including vital signs will be done. Samples of blood and urine will be taken for clinical laboratory and urinalysis. Patients will then undergo a 12-lead ECG test.

A history of side effects with current CBTD as well as laboratory recordings of abnormalities attributable to treatment will also be recorded.

Enrolled subjects will be dosed in a sequential manner, starting with the low dose group (300 mg/day). Safety and tolerability will be monitored closely by an Independent Medical Monitor (IMM) and based on the IMM's assessment that it is safe to proceed to the higher dose (600 mg/day), subsequent subjects will be enrolled into that group. Up to 15 subjects each will be enrolled into either Group A or Group B.

Subjects will stop taking their current CBTDs for 7 days and perform a 24-hour urine collection on Day-7 and report for Day 1 Visit .

Subjects enrolled into Group A will start taking bucillamine tablets orally, three times a day preferably 1hr before or 2hrs after meals in the following sequence; 100 mg (1 tab) in the morning; 100 mg (1 tab) at noon and 100 mg (1 tab) at night. This drug regimen will continue for 7 days. Safety Visits are scheduled on Day 3 and Day 8 (End of Study Visit). Furthermore, on Day 7 a 24-hour urine collection will be performed. Instructions for handling this sample will be provided in a separate manual.

Subjects enrolled into Group B, will start taking bucillamine tablets orally, three times a day preferably 1hr before or 2hrs after meals in the following sequence; 200 mg (2 tabs) in the morning; 200 mg (2 tabs) at noon and 200 mg (2 tabs) at night. This drug regimen will continue for 7 days. Safety Visits are scheduled on Day 3 and Day 8 (End of Study Visit). Furthermore, on Day 7 a 24-hour urine collection will be performed. Instructions for handling this sample will be provided in a separate manual.

After 7 days on the assigned bucillamine dose and after providing the 24-hour urine sample, and after completing the Day 8 safety visit, subjects will undergo a 7 day washout where no CBTDs will be taken. Thereafter, subjects will be allowed to resume their originally prescribed CBTDs under Investigator's supervision.

One week following study drug discontinuation, subjects will return to the clinic for follow-up safety assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects of any gender and of any race ≥18 and ≤80 years of age
2. Subjects with proven cystinuria who are failing their standard drug therapy of tiopronin plus first-line therapy (hydration, alkali and diet restriction) and who meet the following criteria.

   * formed new stones while taking a thiol.
   * had increase in stone size of pre-existing stones while taking a thiol.
   * had a urologic intervention for stones while taking a thiol
3. Subjects must be able to reliably urinate in a collection vessel and measure urine volume
4. Subjects must have documentation of a stable complete blood count (CBC) and urinalysis (UA) in the 6 months prior to date of enrollment
5. Subjects may have a history of but not currently active CNS disorders or symptoms/effects (e.g., headache)
6. Subjects must have adequate organ function, evidenced by the following laboratory results within 30 days prior to enrollment:

   * Absolute neutrophil count >2000 cells/mm
   * Platelet count >140,000 cells/mm3
   * Hemoglobin >11.0 g/dl
   * Albumin ≥2.5 g/dl
   * Total bilirubin ≤1.5 upper limit of normal (ULN)
   * SGOT (aspartate aminotransferase [AST]), SGPT (alanine aminotransferase [ALT]), and alkaline phosphatase (ALP)

     ≤ 2.5 x ULN
   * eGFR >60 ml/min/173m 2 based on Modification of Diet and Renal Disease (MDRD) Study equation which includes the variables of creatinine, age, sex and race
7. Female subject who has been post-menopausal for at least 24 consecutive months, or women who have undergone surgical sterilization, (e.g. hysterectomy, bilateral oophorectomy, tubal ligation or salpingectomy) is eligible without requiring the use of a contraceptive methods described in Inclusion #8
8. For women of childbearing potential and men with partners of childbearing potential, agreement to use a highly effective, non-hormonal form of contraception:

   * Acceptable forms of should include two of the following:

     * Placement of intrauterine device (IUD) or intrauterine system (IUS)
     * Condom with spermicidal foam/gel/film/cream/suppository
     * Diaphragm or cervical/vault caps with spermicidal foam/gel/film/cream/suppository
   * The above contraception is not a requirement in the case of any of the following:

     * Subject is surgically sterilized
     * Subject has had no menstrual period for 12 consecutive months
   * Contraception use should continue for the duration of the study treatment and for at least 3 months after the last dose of study treatment Periodic abstinence (e.g., calendar ovulation, symptom-thermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
9. Subjects must be willing and able to give written informed consent

Exclusion Criteria:

1. Subjects with renal colic
2. Subjects who are scheduled to undergo a surgical procedure
3. Subjects on D-penicillamine (see page 35 for explanation)
4. Subjects with cancer
5. Subjects with acute or chronic infections including HIV, tuberculosis, hepatitis B or hepatitis C
6. Patients with proteinuria ≥30 mg that is confirmed on repeat laboratory assessment within 24 hours
7. Subjects with QTc interval >450 ms
8. A history of, hypokalemia and family history of Long QT syndrome
9. Use of concomitant medications that may prolong QT/QTc interval
10. Patients with significant heart failure and activity impairment (Class III-IV of the New York Heart Association (NYHA)
11. Subjects with serious hepatic disorder (Child-Pugh scores B or C)
12. Subjects with a history of alcohol or substance abuse within the 12 months prior to enrollment
13. Subjects with history of or active blood dyscrasia such as myelosuppression, leukopenia, granulocytopenia, thrombocytopenia, pancytopenia, and aplastic anemia.
14. Subjects with Coagulopathy (regardless if controlled by pharmacotherapy or not)
15. Subjects who have any concomitant illness (including active significant infection) or other finding that, in the opinion of the Investigator, would confound the study data or place the subject at unacceptable risk if the subject were to participate in the study, or that would require frequent adjustments in concomitant medications during the course of the study
16. Use of any investigational drug within 30 days prior to enrollment
17. Subjects currently participating in another research study or anticipated to enroll in such during participation in this study
18. Subjects for whom informed consent cannot be obtained

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Days 0, 2, 3, 7, 8 and + 1 wk post study
  Number, type, and severity of AEs observed by the staff during visits on Days 0 (dosing), 3, 8 and +1 week post-study or volunteered by the subject during telephone follow-up on Days 2 and 7.

SECONDARY OUTCOMES:
Cystine Excretion | Day 0 and Day 8
  Measurement of 24-hr urine cystine excretion.
Cystine Capacity | Day 0 and Day 8
  Measurement of 24-hr urine cystine capacity, i.e., the capacity of a patient's urine to solubilize or precipitate.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - University of Alabama - Department of Urology, Birmingham, Alabama
  - Massachusette General Hospital, Boston, Massachusetts
  - New York University School of Medicine, New York, New York
  - Omega Medical Research, Warwick, Rhode Island
  - University of Wisconsin School of Medicane and Public Health, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No